CLINICAL TRIAL: NCT03430336
Title: Effectiveness and Cost-effectiveness of the Application of an Electronic Medication Management Support System in Patients With Polypharmacy in General Practice (AdAM).
Brief Title: Application for an Electronic Medication Management Support System
Acronym: AdAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BARMER (Other)
Collaborators: Association of Statutory Health Insurance Physicians Westphalia/Lippe, Germany (Unknown); Goethe University (Other); University of Cologne (Other); Ruhr University of Bochum (Other); Bielefeld University (Other); University of Wuppertal (Other)
Responsible Party: Principal Investigator, Christiane Muth, MD, MPH, MD, MPH, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IfA
Record Dates: First submitted 2018-02-06; First posted 2018-02-12 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Polypharmacy
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Masking Description: Due to the character of the intervention, blinding is not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer-assisted medication management (Experimental): Family physician adds, modifies and optimizes medication in patient's with polypharmacy assisted by an user-initiated computerized decision support system (CDSS) which provides drug-therapy relevant information about patients (e.g. diagnoses and treatments) and alerts in case of drug-drug, drug-disease, drug-age interactions to systematically assess the appropriateness of medication:
  * CDSS provides drug-therapy relevant information
  * modification of medication
  * assessment of medication appropriateness
  * medication plan
  * Guidance in medication process
  Interventions: Other: CDSS provides drug-therapy relevant information; Other: Modification of medication; Other: Assessment of medication appropriateness; Other: Medication plan; Other: Guidance in medication process
- Control arm (No Intervention): Patients will receive the usual clinical care based on current clinical practice guidelines during intervention period. After completion of trial, the patients in the control group will be invited to participate after written informed consent to receive the intervention.

INTERVENTIONS:
Other: CDSS provides drug-therapy relevant information — External computerized decision support system (CDSS: RpDoc® eMMa Software, RpDoc® Solutions GmbH, Saarbruecken) provides drug-therapy relevant information about participating patients with polypharmacy on demand to the general practitioners (GPs) such as data about diagnoses and treatments. The information is based on claims data gathered from all health care professionals involved in the care of the patient (e.g. specialized physicians, other GPs, psychotherapists as well as data about hospital stays and prescription data from pharmacies).
  Arms: Computer-assisted medication management
Other: Modification of medication — GPs can add and modify patient's data within the CDSS (e.g. remove drugs which are not taken by the patient anymore, add most recent laboratory findings about kidney function etc.) to enrich and update claims data based information.
  Arms: Computer-assisted medication management
Other: Assessment of medication appropriateness — GPs systematically assess the appropriateness of the medication supported by the CDSS, which will alert in case of drug-drug, drug-disease, and drug-age interactions as well as other inappropriateness, such as prescriptions with regard to incorrect dosage or Dear Doctor letters.
  Arms: Computer-assisted medication management
Other: Medication plan — GPs print out the updated medication plan including also recommendations for medication use and reasons for prescription in lay language (also available in foreign languages for patients with migration background) as well as recommendations on drugs to use / to avoid including over-the-counter drugs (OTC) (optional) and hand it out to the patient.
  Arms: Computer-assisted medication management
Other: Guidance in medication process — GPs receive guidance via the CDSS (e.g. recommendations addressing certain types of medication errors and high risk prescribing, developed by the German Society for Internal Medicine in collaboration with other scientific medical societies).
  Arms: Computer-assisted medication management

SUMMARY:
This study assesses whether an electronic medication management support system improves quality, safety, and cost-effectiveness of the drug therapy in adult patients with polypharmacy compared to usual care during the observation period of 15 months from baseline per practice (from 2017 4th quarter to 2020 3rd quarter).

DETAILED DESCRIPTION:
Title:

Application of an electronic medication management support system.

Objectives:

The aim of the study is to assess the effectiveness of an electronic medication management support system on hospitalization and death, its cost-effectiveness and its effects on the quality and safety of prescribing in patients with polypharmacy.

Methods:

A parallel, cluster-randomised controlled trial will be conducted in about 1,080 general practices located in the Westphalia-Region (Germany), which care for adult patients covered by BARMER health insurance. Per group, 17,200 clustered-randomized patients (about 32 patients per practice) will be included, if they take ≥ 5 long-term prescriptions (at least 2 consecutive quarters).

In the intervention group, family physicians will use an user-initiated clinical decision support system (CDSS) which provides drug-therapy relevant information (e.g. on diagnoses and treatments) and alerts in case of drug-drug, drug-disease and drug-age interactions. Based on that information, the family physician systematically assesses the appropriateness of patient's medication and optimizes it. Patients receive an updated medication plan in their mother's language, if needed.

In the control group, patients continue to receive usual care where there is no access to the CDSS.

The primary outcome is the combined endpoint of all-cause mortality and all-cause hospital admissions after the observation period of 12 quarters or 15 months per practice. The outcome measures will be based on secondary data (i.e. claims data). Primary and secondary outcomes will be measured at patient level. The primary analysis will be performed adhering to the intention-to-treat (ITT) principle.

Amendment (07/04/2020):

The parallel group comparison will be conducted, as planned. However, the design of the primary analysis will be changed into a cluster-randomised stepped wedge design with an open cohort, as the recruitment to the target of N=1,080 practices was not reached. The changes of the design will allow to safe the power of the trial of 80% to detect differences of the combined primary outcome between both groups. The primary outcome as well as the ITT-analysis were not changed. The changes of the design implied the following subsequent adaptations of the protocol:

1. Arms and assigned interventions:

   The GP practices of the intervention group will continue to provide the experimental intervention as described in the experimental arm for the entire time in the trial.

   The GP practices of the control arm (usual care, no intervention) will switch to the experimental arm after five quarters control time and provide the experimental intervention for the remaining time in the trial.
2. Case finding:

   The BARMER creates lists of potentially eligible patients ("Potenzialpatienten") in GP practices participating in the AdAM trial based on the fulfillment of inclusion/exclusion criteria in claims data at each quarter between the first quarter 2018 and the third quarter of 2020.

   Intervention practices receive the lists quarterly from the quarter after randomization and control practices quarterly starting on the date of switch.
3. Informed consent:

The GPs in practices of the experimental arm (either they were randomized and assigned as intervention practices at the beginning of the trial or they switch after the end of five quarters control time) invite potentially eligible patients from the lists and ask for a written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with polypharmacy (5 or more drugs taken for at least two quarters).
* Informed consent.

Exclusion Criteria:

* Incapacitated patients without legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of all-cause mortality and all-cause hospital admissions | Observation period of 15 months per practice
  The primary outcome is the combined endpoint of all-cause mortality and all-cause hospital admissions (including night- and day-only admissions) in patients with polypharmacy.

SECONDARY OUTCOMES:
Number of potential inappropriate prescriptions | Observation period of 15 months per practice
  Number of potential inappropriate prescriptions: to ascertain whether the complex intervention improves the appropriateness of prescriptions (high-risk prescriptions) in patients with polypharmacy.
All-cause hospital admissions | Observation period of 15 months per practice (quarterly)
  All-cause hospital admissions: to evaluate whether the complex intervention reduces all-cause hospital admissions (including day- or night-only admissions) (number and duration) in patients with polypharmacy.
All-cause mortality | Observation period of 15 months per practice (quarterly)
  All-cause mortality: to assess whether the complex intervention reduces all-cause mortality in patients with polypharmacy.

OTHER OUTCOMES:
Cost Effectiveness | Observation period of 15 months per practice
  Cost-effectiveness of the intervention will be measured by the incremental cost-effectiveness ratio (ICER), which is expressed as the ratio of the difference in overall costs between the control and the intervention group and the difference in effects between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Kellermann-Mühlhoff, Study Director — BARMER Health Insurance
Locations (2):
- Germany (2):
  - Association of Statutory Health Insurance Physicians Westphalia/Lippe, Dortmund
  - BARMER Health Insurance, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piotrowski A, Coenen J, Rupietta C, Basten J, Muth C, Soling S, Zimmer V, Karbach U, Kellermann-Muhlhoff P, Koberlein-Neu J; AdAM study group. Factors facilitating the implementation of a clinical decision support system in primary care practices: a fuzzy set qualitative comparative analysis. BMC Health Serv Res. 2023 Oct 26;23(1):1161. doi: 10.1186/s12913-023-10156-9. PMID 37884934
- [Derived] Freund J, Piotrowski A, Buhrmann L, Oehler C, Titzler I, Netter AL, Potthoff S, Ebert DD, Finch T, Koberlein-Neu J, Etzelmuller A. Validation of the German Normalisation Process Theory Measure G-NoMAD: translation, adaptation, and pilot testing. Implement Sci Commun. 2023 Oct 16;4(1):126. doi: 10.1186/s43058-023-00505-4. PMID 37845776
- [Derived] Soling S, Demirer I, Koberlein-Neu J, Hower KI, Muller BS, Pfaff H, Karbach U; AdAM Study Group. Complex implementation mechanisms in primary care: do physicians' beliefs about the effectiveness of innovation play a mediating role? Applying a realist inquiry and structural equation modeling approach in a formative evaluation study. BMC Prim Care. 2023 Jun 27;24(1):131. doi: 10.1186/s12875-023-02081-x. PMID 37369994
- [Derived] Muller BS, Klaassen-Mielke R, Gonzalez-Gonzalez AI, Grandt D, Hammerschmidt R, Koberlein-Neu J, Kellermann-Muhlhoff P, Trampisch HJ, Beckmann T, Duvel L, Surmann B, Flaig B, Ihle P, Soling S, Grandt S, Dinh TS, Piotrowski A, Meyer I, Karbach U, Harder S, Perera R, Glasziou P, Pfaff H, Greiner W, Gerlach FM, Timmesfeld N, Muth C; AdAM study group. Effectiveness of the application of an electronic medication management support system in patients with polypharmacy in general practice: a study protocol of cluster-randomised controlled trial (AdAM). BMJ Open. 2021 Sep 28;11(9):e048191. doi: 10.1136/bmjopen-2020-048191. PMID 34588245
- [Derived] Brunn R, Muller BS, Flaig B, Kellermann-Muhlhoff P, Karbach U, Soling S, Muth C, van den Akker M; AdAM Study consortium. "I must, and I can live with that": a thematic analysis of patients' perspectives on polypharmacy and a digital decision support system for GPs. BMC Fam Pract. 2021 Aug 21;22(1):168. doi: 10.1186/s12875-021-01517-6. PMID 34418964
- [Derived] Soling S, Koberlein-Neu J, Muller BS, Dinh TS, Muth C, Pfaff H, Karbach U; AdAM Study Group. From sensitization to adoption? A qualitative study of the implementation of a digitally supported intervention for clinical decision making in polypharmacy. Implement Sci. 2020 Sep 21;15(1):82. doi: 10.1186/s13012-020-01043-6. PMID 32958010